CLINICAL TRIAL: NCT05365308
Title: EHR-based Patient Identification and Panel Management of Patients With Iron Deficiency Anemia, a Pragmatic Primary Care Physician Randomized Trial of a Quality Improvement Method
Brief Title: EHR-based Patient Identification and Panel Management of Patients With Iron Deficiency Anemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Stephen Persell, MD, MPH, Professor of Medicine, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STU00213747
Record Dates: First submitted 2022-04-14; First posted 2022-05-09 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Iron-deficiency Anemia
MeSH Terms: conditions — Anemia, Iron-Deficiency

STUDY DESIGN:
Intervention Model Description: Stratified physician-randomized controlled quality improvement intervention study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Quality Improvement tools (Experimental): Quality improvement tools including: computer-assisted identification of iron deficiency anemia patients with an EHR registry, facilitated GI referral, an EHR tool for documentation, and physician education.
  Interventions: Behavioral: Clinical supports
- Control: usual care (No Intervention): Physicians will be notified at the start of the study that 120 days after the study start they will receive access to the quality improvement tools available to the intervention group.

INTERVENTIONS:
Behavioral: Clinical supports — Quality improvement tools for iron deficiency anemia that include computer-assisted identification, an EHR registry, facilitated GI referral, an EHR tool for documentation, and physician education
  Arms: Intervention: Quality Improvement tools

SUMMARY:
The objective is to determine if a set of clinical supports that includes computer-assisted identification, an EHR registry, facilitated GI referral, and an EHR tool for documentation improves the timely referral and completion of bidirectional endoscopy in men aged 18 years and older and women aged 40 years and older with iron deficiency anemia.

ELIGIBILITY:
Inclusion Criteria:

Northwestern Medical Group primary care physician (internal medicine, family medicine or geriatrics)

Exclusion Criteria:

No primary care office practice within Northwestern Medical Group

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-06-28 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
Bidirectional endoscopy completed | 120 days
  Completion of upper and lower endoscopy, assessed using automated queries of the Northwestern Medicine Enterprise Data Warehouse occurring within the three years prior to the study start date and the 120 days following the study start date.
  Specificially, presence of one or more terms for a completed procedure from the code set for Espohagoduodenoscopy/Upper Endoscopy and one or more terms from the code set for Colonoscopy within the indicated time frame constitutes completion of the measure.
  Note:the investigators use a three-year look back because eligible patients may have completed either upper or lower endoscopy previously and only require one form of endoscopy during the study period.

SECONDARY OUTCOMES:
Endoscopy completed or scheduled | 120 days
  Discrete evidence in the EHR that endoscopy has been completed or scheduled on or after the study start date.
  Specificially, presence in the Northwestern Medicine EHR of a completed or future scheduled procedure for one or more terms from the code set for Espohagoduodenoscopy/Upper Endoscopy or one or more terms from the code set for Colonoscopy within the indicated time frame constitutes completion of the measure.
  Note:the investigators use a three-year look back because eligible patients may have completed either upper or lower endoscopy previously and only require one form of endoscopy during the study period.
Gastroenterology consultation completed | 120 days
  Completion of a consultation with gastroenterology (in person or telehealth) on or after the study start date
  Specificially, this outcome is indicated by the presence in the Northwestern Medicine EHR of a completed office visit or telehealth visit with a physician, physician assistant or advance practice nurse in the within the specialty department of gastroenterology.
GI referral provided or completed | 120 days
  Receipt of a referral to gastroenterology or completion of a consultation with gastroenterology
  Specificially, this outcome is indicated by the presence in the Northwestern Medicine EHR of a completed office visit or telehealth visit with a physician, physician assistant or advance practice nurse in the within the specialty department of gastroenterology or the presence of a signed order for a gastroenterology referral or an endoscopy referral.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Northwestern University, Division of General Internal Medicine, Chicago, Illinois
  - Stephen D Persell, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No
No data sharing plan.

REFERENCES:
- [Derived] Priyanath Gupta A, Patel D, Lee JY, Volpentesta M, Schachter M, Persell SD. Health information technology tools to accelerate gastrointestinal evaluation in patients with iron deficiency anaemia: a cluster randomised controlled trial. BMJ Open Qual. 2024 Apr 15;13(2):e002565. doi: 10.1136/bmjoq-2023-002565. PMID 38626940